CLINICAL TRIAL: NCT05804331
Title: The Australia and New Zealand Multicentre Upper Gastrointestinal Endoscopic Tissue Resection Study
Acronym: ANZ UGI
Status: Recruiting | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Director of Endoscopy, Western Sydney Local Health District
Other Study IDs: 2022/PID02709
Record Dates: First submitted 2023-03-12; First posted 2023-04-07 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Cancer of Stomach; Oesophageal Cancer; Gastric Cancer; Gastric Adenocarcinoma; GI Cancer; GIST; Neuroendocrine Tumors; Gastric Neoplasm; Esophageal Neoplasms
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Gastrointestinal Neoplasms; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with Gastrointestinal neoplasm: Pt referred for resection of gastrointestinal neoplasm. Observational data collected from endoscopic submucosal dissection (ESD), submucosal-tunnelling endoscopic resection (STER) or endoscopic full-thickness resection (EFTR) of gastrointestinal neoplasm

SUMMARY:
To determine the long term outcomes of Endoscopic Submucosal Dissection (ESD), Endoscopic Full Thickness Resection (EFTR) and Submucosal-Tunnelling Endoscopic Resection (STER) for upper gastrointestinal neoplastic lesions

DETAILED DESCRIPTION:
To collect prospective observational data on patients undergoing ESD, EFTR or STER for UGI neoplastic lesions

* Lesion characteristics including histology
* Procedural outcomes
* Safety Outcomes
* Efficacy outcomes

ELIGIBILITY:
Inclusion Criteria:

* UGI neoplastic lesions > 10mm

  * Lesions for ESD limited to the mucosal and/or submucosal layer OR
  * Lesions for EFTR limited to the muscularis propria layer OR
  * Lesions for STER limited to the submucosal and/or muscularis propria layer
* Aged 18 years or older

Exclusion Criteria:

* Age less than 18
* Unable to give informed consent
* Pregnant or lactating patients
* Patients with bleeding diathesis or who cannot discontinue ADP blockers (e.g. clopidogrel, prasugrel) or antithrombotics (e.g. warfarin, dabigatran) periprocedurally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to tertiary centre for endoscopic resection of gastrointestinal neoplasm
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2028-03-14 (Estimated); Study Completion 2028-09-14 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of endoscopic resection of UGI neoplastic lesions: completeness of resection | 2 weeks
  Determined based on clear margins in histology review
Safety: intra and post procedural; bleeding; perforation; anaesthetic | 30 day
  Intraprocedural bleeding, clinically significant post-polypectomy bleeding, deep mural injury, post polypectomy coagulation syndrome
Long term outcomes: recurrent and residual disease | 3 years
  Determined at subsequent procedures

SECONDARY OUTCOMES:
Endoscopic sessions, procedure time (in minutes) and overall time (in weeks) needed to achieve the primary objectives | 6 months
  Determined after follow up procedure to confirm no recurrence
Need for more than one endoscopic therapy | 3 years
  Determined after follow up procedures
Need for surgery | 2 months
  Determined after follow up procedures, histological review
Post ESD, EFTR, STER defect features | 1 day
  Determined after complete resection
Patient interviews/questionnaires | 3 years
  Determined after follow up procedures

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, Principal Investigator — WSLHD
Locations (1):
- Westmead Hospital, Sydney, New South Wales, Australia